CLINICAL TRIAL: NCT04472052
Title: Incidence of Perforated Appendicitis in Times of Corona Crisis
Brief Title: Frequency of Perforated Appendicitis in Times of COVID-19
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: AZ: 324/2020BO2
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Perforated Appendicitis; Covid19
Keywords: acute appendicitis, COVID-19
MeSH Terms: conditions — Appendicitis; COVID-19 | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Appendectomy: Patients who required appendectomy for suspected acute appendicitis
  Interventions: Other: appendectomy

INTERVENTIONS:
Other: appendectomy — Surgical standard treatment for acute appendicitis All patients receive preoperative single-shot antibiosis, usually 2000 mg cefotaxime combined 500 mg metronidazole. Appendectomy is performed usually within 24 h of admission in patients with acute appendicitis. The laparoscopic appendectomy using the 3-trocar technique represents the surgical standard. In uncomplicated or non-perforated appendicitis, drainage is generally not required. Wounds are closed intra-cutaneous with absorbable sutures. Patients without postoperative complications are discharged home two days after surgery.

SUMMARY:
Appendicitis is one of the most common clinical conditions in general surgery. The diagnosis is usually made from clinical examination, imaging (sonography or CT) and laboratory parameters. The laparoscopic appendectomy without drainage has established as the gold standard. Patients usually leave the hospital two days after surgery.

In times of corona crisis, patients are unsure to visit the hospital because of fear of infection with SARS-CoV-2. A higher incidence of perforated appendicitis could be an indicator for fear-related delay of going to the hospital.

Methods: Investigators performed a retrospective analysis on the incidence of perforated appendicitis in a 10-week interval (mid-March to end of May) of the years 2018, 2019 and 2020 to evaluate possible changes in times of corona crisis. Intraoperative findings, procedures, complications and the length of hospital stay were considered.

DETAILED DESCRIPTION:
The local ethics committee of the University Hospital of Tübingen, Germany, approved this study (AZ: 324/2020BO2). All patients treated for acute appendicitis in a ten week period from 16th of March to 31th of May in 2018, 2019 and 2020 were considered for the study. Investigators analysed the frequency of perforated appendicitis in the periods indicated. Informed consent was obtained from all individual participants. Patient's records as well as database were analyzed for therapy specific items.

Definition Perforation: Perforated appendicitis was defined as described perforation in the surgical or pathological results.

Delay between onset of symptoms and first presentation at the hospital: Patient's records were proved for self-declaration about the start of symptoms

ELIGIBILITY:
Inclusion Criteria:

* patients with acute appendicitis older than 16 years
* appendectomy in time frame 16th of march to 30th of May in the Years 2018, 2019 and 2020

Exclusion Criteria:

* patients with acute appendicitis younger than 16 years
* appendectomy not in the named time frames

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
rate of perforated appendicitis | 10 weeks from 16th of March to 31th of May

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
Researchers could send a request for the IPD to the investigators and will receive the required data.